CLINICAL TRIAL: NCT01746212
Title: Outcomes of Patients With Lumbar Degenerative Disc Disease Treated Operatively With an Anterior-Only Approach Using InQu Bone Graft Extender and Substitute
Brief Title: Outcomes of Degenerative Disc Disease Patients Treated With an Anterior-Only Fusion Using InQu Bone Graft
Acronym: InQu
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kansas Joint and Spine Institute (Network)
Collaborators: National Center of Innovation for Biomaterials in Orthopaedic Research (Unknown); ISTO Technologies, Inc. (Industry)
Responsible Party: Principal Investigator, Mark Camden Whitaker, Principal Investigator, Kansas Joint and Spine Institute
Other Study IDs: InQu ALIF
Record Dates: First submitted 2012-12-03; First posted 2012-12-10 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Degenerative Disc Disease
Keywords: Degenerative Disc Disease; InQu Bone Graft Extender and Substitute; Anterior Lumbar Interbody Fusion; Oswestry Disability Index; Visual Analog Scale; Stand-alone ALIF; Bone Marrow Aspirate Concentrate; Fusion rate; Disc Height; Mean Optical Density; Integrated Optical Density
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Degenerative Disc Disease: Patients diagnosed with degenerative disc disease, meeting all eligibility requirements (please refer to inclusion/exclusion criteria), will be asked to participate in this study. A one-level or two-level anterior lumbar interbody fusion surgery using InQu Bone Graft Extender and Substitute, mixed with BMAC (bone marrow aspirate concentrate) as autograft, with Synthes Spinal Instrumentation will be recommended to the patient. If patients elect to proceed with surgery using the prescribed surgical components, they will be offered enrollment into the study. If the patient opts to use a different bone graft, or other spinal instrumentation, then the patient will not meet all inclusion criteria and will not be offered the opportunity to enroll in this study.
  Interventions: Procedure: One-level or two-level anterior lumbar interbody fusion; Biological: InQu Bone Graft Extender and Substitute mixed with BMAC; Device: Synthes Spinal Instrumentation

INTERVENTIONS:
Procedure: One-level or two-level anterior lumbar interbody fusion — Patients electing to receive a one-level or two-level, anterior approach only (incision through the front), lumbar interbody fusion in order to treat degenerative disc disease (at one or two levels in the spine), and meeting all other inclusion criteria, are eligible for enrollment into the study.
  Other Names: ALIF
Biological: InQu Bone Graft Extender and Substitute mixed with BMAC — Surgeries utilizing InQu Bone Graft Extender and Substitute during the anterior lumbar interbody fusion surgical procedure will be elected for inclusion. InQu will be mixed with BMAC (bone marrow aspirate concentrate), which will be prepared using the SmartPRep2 centrifuge. Patients opting to use a grafting alternative will not meet inclusion criteria, and will not be eligible to enroll in this study.
  Other Names: InQu; BMAC; SmartPRep2 centrifuge
Device: Synthes Spinal Instrumentation — Synthes Spinal Instrumentation will be used during surgery as spinal stabilization.
  Other Names: ATB Plate; Peek Cage; SynFix-LR

SUMMARY:
The purpose of this study is to report the radiographic, clinical, and functional outcomes of a consecutive series of patients diagnosed with single or bilateral degenerative disc disease between L4 and S1, that have been treated with an anterior lumbar interbody fusion (ALIF), anterior only surgical approach, and InQu Bone Graft Extender and Substitute for bony fusion and instrumentation.

Patients that decide to undergo an Anterior Lumbar Interbody Fusion (ALIF) surgery [a surgical procedure that joins two or more lumbar vertebrae (small bones of the spine) together into one solid bony structure by approaching the spine through the abdomen (front of the body) and placing a bone graft in between the vertebral bodies where the disc usually lies], are invited to participate in an orthopaedic research study.

This study will compare patients that have been treated with an anterior lumbar interbody fusion using InQu Bone Graft Extender & Substitute to published data for a stand alone spinal fusion surgery, where InFuse bone graft is placed between the transverse processes [small bony projections off the right and left side of each bone in your spine] of the affected vertebrae.

X-rays, daily activities, and how patients are doing will be evaluated at specific time points during this study.

The hypothesis of this study is that patients diagnosed with degenerative disc disease treated with an anterior lumbar interbody fusion, anterior only surgical approach (incision through the abdomen), using InQu Bone Graft Extender and Substitute and instrumented fixation have comparable radiographic (x-rays), functional (daily activities), and clinical (how the patient is doing) outcomes when compared to published data for use of InFuse in stand-alone fusion.

DETAILED DESCRIPTION:
This is a prospective, observational study; evaluating outcomes of patients that have elected to receive surgical intervention in order to treat degenerative disc disease. In order to be eligible for enrollment into this study, patients have already elected to be treated with an anterior lumbar interbody fusion, an anterior only approach for single or bi-level degenerative disc disease between L4 and S1 with instrumented fusion, using a combination of InQu Bone Graft Extender and Substitute, local bone, and Bone Marrow Aspirate Concentrate (BMAC) to promote bony fusion. Only after the patient and physician determine the surgical procedure, can the patient be eligible for enrollment. A consecutive series of 60 patients will be offered enrollment if all inclusion/exclusion criteria are met.

Data will be collected by chart review to include pre-operative, surgical, functional, post-operative, and radiographic imaging charted data, collected as part of the routine clinical visit, and standard of care.

Follow-up data will include newly charted clinical, functional, and radiographic imaging data, including dynamic x-rays and CT scans to be obtained prospectively at a minimum of one (1) year post-operatively. During the routine post-surgical visits, patient pain outcomes are measured using the Visual Analog Scale (VAS) for back and leg pain, function is measured by the Oswestry Disability Index (ODI) and Short Form-12 Version 2 (SF-12 Version 2 Health Survey). A physician investigator will also perform routine clinical evaluations.

The patients will undergo standard radiographic procedures to obtain x-rays (including lateral, anterior-posterior, and dynamic flexion/extension) as part of the standard of care. A CT scan will be performed for research purposes as indicated in the protocol follow-up procedure. X-rays and CT scans will be evaluated by an independent radiologist and a physician investigator to determine anterior fusion status and the status of the anterior hardware constructs.

The National Center of Innovation for Biomaterials in Orthopaedic Research and Medical Metric, Inc. will assist with imaging analysis of x-rays and CTs.

ISTO Technologies, Inc. will be providing a grant to cover costs associated with the research components of this study.

ELIGIBILITY:
Inclusion Criteria: Patients are eligible for this study if the following criteria are all met.

* Patient will be surgically treated with an anterior lumbar interbody fusion, anterior only approach by one of the listed physician investigators
* Must have had a structural problem potentially amendable to primary fusion at one or two levels
* InQu Bone Graft Extender and Substitute will be used in the surgery
* Had failed conservative care for longer than three (3) months
* Had no psychological contraindications for surgery
* Aged 18 to 70 years of age at the time of surgery

Exclusion Criteria: Patients are ineligible for this study if any one of the following criteria apply.

* Patients that will not be surgically treated with an anterior lumbar interbody fusion, anterior only approach by one of the physician investigators
* InQu Bone Graft Extender and Substitute will not be used in the surgery
* Patient carries any one of the following diagnoses: spinal stenosis requiring decompression, isthmic spondylolisthesis, degenerative spondylolisthesis greater than three (3) millimeters, three or more degenerative levels, major deformity, have had a previous lumbar fusion, or if they have had a previous infection or tumor
* Individuals that can not provide consent for themselves
* Patients requiring revision surgery
* Aged younger than 18 or older than 70 at the time of surgery
* Patients will be excluded from participating in the study if, in the investigators' opinion, they will be unable to comply with study procedures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Target population included adult patients from the normal patient population seen at Kansas Joint and Spine Institute, currently also known as Kansas Spine Specialists, that have the ability to provide informed consent without assistance. Each patient that is qualified for an anterior lumbar interbody fusion, with an anterior only approach, will be offered the InQu Bone Graft Extender and Substitute as the bone graft the investigator will use in surgery. Patients that proceed with surgical intervention, and that meet all inclusion/exclusion criteria, will be offered enrollment into the study.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-12; Primary Completion 2015-03 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Evidence of successful radiographic fusion at 1-year post-operative | 12-months post-operative
  X-rays and CTs will be analyzed for fusion based on the following criteria:
  1. Bridging trabecular bone connecting the two vertebral bodies either through the dowels or around the dowels as evaluated by thin-cut CT scans and radiographs;
  2. No angular motion of 5 degrees or more on dynamic plain radiographs;
  3. No sagittal translation of more than 3 mm on dynamic plain radiographs; and
  4. No radiolucencies that involve more than half of the interfaces between the dowels and the host vertebral end plates.
  Criteria is based on the Burkus, Transfelt, et. al study titled "Clinical and Radiographic Outcomes of Anterior Lumbar Interbody Fusion Using Recombinant Human Bone Morphogenetic Protein-2."

SECONDARY OUTCOMES:
Improvement in Oswestry Disability Index Score (1-year) | Change from baseline to 12-months post-operative
  Change in ODI and between baseline and 1-year post-operative, anticipating improvement in ODI score (i.e. from baseline to 12-months post-operative, scores should decrease).
Improvement in Oswestry Disability Index Scores (2-years) | Change from baseline to 24-month post-operative
  Change in ODI and between baseline and 2-year post-operative, anticipating improvement in ODI score (i.e. from baseline to 24-months post-operative, scores should decrease).
Improvement in Visual Analog Scale Scores (1-year) | Change from baseline to 12-months post-operative
  Change in VAS and between baseline and 1-year post-operative, anticipating improvement in VAS score (i.e. from baseline to 12-months post-operative, scores should decrease).
Improvement in Visual Analog Scale Scores (2-years) | Change from baseline to 24-months post-operative
  Change in VAS and between baseline and 2-year post-operative, anticipating improvement in VAS score (i.e. from baseline to 24-months post-operative, scores should decrease).

OTHER OUTCOMES:
Surgical Outcomes | At time of surgery
  Estimated blood loss, Operative time, Hospital stay
Radiographic Measurements at 6-months post-operative | Change from baseline to 6-months post-operative
  Evaluation of Disc Height, Mean Optical Density, and Integrated Optical Density
Radiographic Measurements at 12-months post-operative | Change from baseline to 12-months post-operative
  Evaluation of Disc Height, Mean Optical Density, and Integrated Optical Density
Radiographic Measurements at 18-months post-operative | Change from baseline to 18-months post-operative
  Evaluation of Disc Height, Mean Optical Density, and Integrated Optical Density
Radiographic Measurements at 24-months post-operative | Change from baseline to 24-months post-operative
  Evaluation of Disc Height, Mean Optical Density, and Integrated Optical Density

CONTACTS AND LOCATIONS:
Overall Officials: Mark C Whitaker, MD, Principal Investigator — Kansas Joint and Spine Institute
Locations (2):
- United States (2):
  - Kansas Joint and Spine Institute, Wichita, Kansas
  - National Center of Innovation for Biomaterials in Orthopaedic Research, Wichita, Kansas